CLINICAL TRIAL: NCT04762875
Title: A Phase II Study Evaluating the Safety and Efficacy of MGTA-145 in Combination With Plerixafor for the Mobilization and Transplantation of HLA-Matched Donor Hematopoietic Stem Cells in Recipients With Hematological Malignancies
Brief Title: MGTA-145 + Plerixafor in the Mobilization of HSCs for Allogeneic Transplant in Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was voluntarily terminated due to a business decision not to proceed and not due to any safety issue
Sponsor: Ensoma (Industry)
Collaborators: National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 145-ADS-202
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Related Donors Donating PBSC to a Family Member; Healthy Donors; Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single dose MGTA-145 plus plerixafor followed by apheresis (Experimental): MGTA-145 in combination with plerixafor followed by apheresis on one or two consecutive days
  Interventions: Biological: MGTA-145; Biological: Plerixafor

INTERVENTIONS:
Biological: MGTA-145 — MGTA-145 will be be administered as an IV infusion
Biological: Plerixafor — 240 µg/kg subcutaneously
  Other Names: Mozobil

SUMMARY:
This research study tests a new medicine for mobilizing stem cells so they can be collected and used for allogeneic stem cell transplant for treatment of hematological malignancies. MGTA-145, the new medicine, will be given with plerixafor.

DETAILED DESCRIPTION:
This is a Phase II, open-label, multicenter, prospective study of MGTA-145 + plerixafor mobilized HLA-matched sibling and matched unrelated donor allografts for myeloablative hematopoietic stem cell transplantation (HSCT) in recipients with hematological malignancies. Donors will undergo 1 or 2 days of mobilization and apheresis.

ELIGIBILITY:
Inclusion Criteria:

Donor Inclusion Criteria:

* Donor medical suitability and eligibility will be determined following Institution or NMDP/Be The Match standards
* Age 18-65 years old at the time of signing informed consent
* 8/8 (HLA- A, B, C, and DRB1) HLA-matched sibling or volunteer unrelated donor
* Fulfill Institution or NMDP/Be The Match criteria to serve as a mobilized blood cell donor
* Serum creatinine < 1.5 x institution upper limit of normal (ULN) or estimated creatinine clearance (CRCL) > 50 mL/min using the Modification of Diet in Renal Disease Study (MDRD) equation or similar method

Recipient Inclusion Criteria:

* At least 18 years old at the time of signing informed consent
* Has an available 8/8 (HLA- A, B, C, and DRB1) HLA-matched sibling or volunteer unrelated donor willing to donate peripheral blood stem cells (PBSC) for transplant
* Fulfill additional individual Transplant Center Criteria for transplant beyond NMDP/Be The Match criteria
* One of the following diagnoses:

  * Acute myelogenous leukemia (AML) in 1st remission or beyond with ≤ 5% marrow blasts and no circulating blasts. Documentation of bone marrow assessment will be accepted within 45 days prior to the date of consent.
  * Acute lymphoblastic leukemia (ALL) in 1st remission or beyond with ≤ 5% marrow blasts and no circulating blasts. Documentation of bone marrow assessment will be accepted within 45 days prior to the date of consent.
  * Patients with myelodysplasia (MDS) with no circulating blasts and with less than 10% blasts in the bone marrow (higher blast percentage allowed in MDS due to lack of differences in outcomes with < 5% or 5-10% blasts in MDS). Documentation of bone marrow assessment will be accepted within 45 days prior to the date of consent.
* Cardiac function: Left ventricular ejection fraction at least 45% based on most recent echocardiogram or MUGA results obtained via standard of care
* Estimated creatinine clearance acceptable per local institutional guidelines
* Pulmonary function: diffusing capacity of the lungs for carbon monoxide (DLCO) corrected for hemoglobin at least 50% and forced expiratory volume in first second (FEV1) predicted at least 50% based on most recent DLCO results obtained via standard of care
* Liver function acceptable per local institutional guidelines
* Karnofsky performance status (KPS) of 70% or greater
* Hematopoietic Cell Transplantation-Comorbidity Index (HCT-CI) score of 4 or less

Exclusion Criteria:

Donor Exclusion Criteria:

* Donor unwilling or unable to give informed consent, or unable to comply with the protocol including required follow-up and testing
* Donor already enrolled on another investigational agent study
* Pregnant or breastfeeding females, sexually active female and male donors not willing or able to use adequate contraception, or males who do not agree to refrain from donating sperm, from the time of consent through 3 months after treatment with MGTA-145 + plerixafor

Recipient Exclusion Criteria:

* Subject unwilling or unable to give informed consent, or unable to comply with the protocol including required follow-up and testing
* Subject whose donor does not meet the eligibility criteria and is a screen fail
* Subjects with a prior allogeneic transplant
* Subjects with active, uncontrolled infection at the time of the transplant preparative regimen
* Pregnant or breastfeeding females, sexually active female or male subjects not willing or able to use adequate contraception, or males who do not agree to refrain from donating sperm, from the time of consent through 3 months after PBSC infusion
* Subjects with clinical evidence of active Central Nervous System (CNS) tumor involvement as evidenced by documented disease on examination of spinal fluid or MRI within 45 days of start of conditioning
* A condition, which, in the opinion of the clinical investigator, would interfere with the evaluation of primary and secondary endpoints
* Planned treatment with a new investigational agent from the time of transplant through 30 days post-transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Devine, MD, Study Chair — National Marrow Donor Program
Locations (8):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Health Care, Stanford, California
  - Emory University Hospital, Atlanta, Georgia
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ohio State Medical Center, James Cancer Center, Columbus, Ohio
  - M.D. Anderson Cancer Center, Houston, Texas
  - Be The Match Collection Center Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis: Donor population
  MGTA-145 in combination with plerixafor followed by apheresis on one or two consecutive days
  MGTA-145: MGTA-145 will be be administered as an IV infusion
  Plerixafor: 240 µg/kg subcutaneously
- Subjects Transplanted With Plerixafor + MGTA-145 Mobilized Product: Transplant recipient after donors mobilized with single-dose MGTA-145 plus plerixafor
Period: Overall Study
Arm/Group | Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis | Subjects Transplanted With Plerixafor + MGTA-145 Mobilized Product
Started | 4 | 3
Completed | 3 | 0
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis | Subjects Transplanted With Plerixafor + MGTA-145 Mobilized Product | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Median (Full Range); unit: years] | 44 [35 to 63] | 61 [26 to 63] | 45 [26 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Weight [Median (Full Range); unit: kg] | 73.7 [66.7 to 91.8] | 81 [55 to 97] | 77 [55 to 97]

OUTCOME MEASURES:

1. Primary Outcome: HSC Yield in Apheresis Product
Description: Number of subjects with adequate number of hematopoietic stem cells (≥ 2.0 x 10^6 CD34+ cells/kg) in one apheresis setting.
Time Frame: Up to 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis
Number analyzed (Participants) | 4
Participants | 2

2. Secondary Outcome: HSC Yield in Apheresis Product
Description: To determine the proportion of donors whose cells can be successfully mobilized and collected with a target CD34+ cell dose of at least 4.0 x 10^6 CD34+ cells/kg actual recipient weight in one apheresis collection
Time Frame: Up to 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis
Number analyzed (Participants) | 4
Participants | 2

3. Secondary Outcome: Adverse Events Experienced by Donors
Description: To ascertain the incidence of adverse events (AEs) before and during apheresis experienced by donors receiving MGTA-145 + plerixafor
Time Frame: Baseline though day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis
Number analyzed (Participants) | 4
Participants | 4

4. Secondary Outcome: Graft Durability
Description: The proportion of participants with primary and secondary graft failure after transplantation of hematopoietic cells mobilized with MGTA-145 + plerixafor
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis
Number analyzed (Participants) | 3
Participants | 0

5. Secondary Outcome: Graft-versus Host Disease (GVHD)
Description: To determine the incidence of acute and chronic graft versus host disease (GVHD) after transplantation of hematopoietic cells mobilized with MGTA-145 + plerixafor
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis
Number analyzed (Participants) | 3
Participants | 0

6. Secondary Outcome: Treatment-related Mortality
Description: To determine the proportion of treatment-related mortality and disease relapse/progression after transplantation of hematopoietic cells mobilized with MGTA-145 + plerixafor
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis
Number analyzed (Participants) | 3
Participants | 0

7. Secondary Outcome: Overall Survival
Description: To determine the probability of overall survival after transplantation of hematopoietic cells mobilized with MGTA-145 + plerixafor
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis | Subjects Transplanted With Plerixafor + MGTA-145 Mobilized Product
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/3
Other Adverse Events (participants affected / at risk) | 4/4 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis (N=4) | Subjects Transplanted With Plerixafor + MGTA-145 Mobilized Product (N=3)
Secondary Graft Loss (Blood and lymphatic system disorders) | 0 | 1
Upper GI Hemorrhage (Gastrointestinal disorders) | 0 | 1
Aspergillus pneumonia (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Dose MGTA-145 Plus Plerixafor Followed by Apheresis (N=4) | Subjects Transplanted With Plerixafor + MGTA-145 Mobilized Product (N=3)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain - arm (General disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Platelet count decreased (Investigations) | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 — Arm cramping
Dysesthesia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Mild face tingling (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT04762875/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT04762875/SAP_001.pdf